CLINICAL TRIAL: NCT00001037
Title: A Phase I, Multicenter, Clinical Trial to Evaluate the Safety and Immunogenicity of Vaccinia-Derived MN HIV-1 Recombinant Envelope Glycoprotein (rgp160) of Human Immunodeficiency Virus at Two Different Vaccination Schedules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: AVEG 013A; 10559 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)

SUMMARY:
To determine the safety and immunogenicity of 200 mcg MN rgp160 vaccine (Immuno-AG) versus placebo, administered on two immunization schedules to healthy volunteers. Per 06/15/94 amendment, to determine the safety and immunogenicity of 800 versus 200 mcg given as a fourth immunization at 9 or 11 months after the third injection (i.e., at month 17).

A gp160 vaccine developed from the IIIB strain of HIV-1 has been found to be safe and immunogenic in healthy adults. Since the MN strain of HIV-1 is representative of a larger proportion of HIV-1 isolates in the United States than is the IIIB strain, evaluation of a gp160 vaccine derived from the MN strain is important.

DETAILED DESCRIPTION:
A gp160 vaccine developed from the IIIB strain of HIV-1 has been found to be safe and immunogenic in healthy adults. Since the MN strain of HIV-1 is representative of a larger proportion of HIV-1 isolates in the United States than is the IIIB strain, evaluation of a gp160 vaccine derived from the MN strain is important.

Volunteers are randomized to receive 200 mcg MN rgp160 or placebo at months 0, 1, and 6 or at months 0, 2, and 8. For each immunization schedule, ten volunteers receive vaccine and two volunteers receive placebo. Per amendment, volunteers receive a fourth immunization of 800 or 200 mcg (or placebo) at 9 or 11 months after the third injection (i.e., at month 17) and are followed for 6 months afterward.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative test for HIV by ELISA within 6 weeks prior to immunization.
* CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrate.
* No history of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppresssive medications.

Exclusion Criteria

Co-existing Condition:

Subjects with the following conditions are excluded:

* Positive for hepatitis B surface antigen.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance.
* Active syphilis (NOTE: If serology is documented to be a false positive or due to a remote (> 6 months) infection, subject is eligible).
* Active tuberculosis (NOTE: Subjects with a positive PPD and normal x-ray showing no evidence of TB and who do not require INH therapy are eligible).

Subjects with the following prior conditions are excluded:

* History of anaphylaxis or other serious adverse reactions to vaccines.

Prior Medication:

Excluded:

* Prior HIV vaccines.
* Live attenuated vaccines within the past 60 days. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) do not exclude but should be administered at least 2 weeks prior to HIV immunizations.
* Experimental agents within the past 30 days.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Higher risk behavior for HIV infection as determined by screening questionnaire, including:

* History of injection drug use within 12 months prior to study entry.
* Higher or intermediate risk sexual behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Study Completion 1995-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gorse G, Study Chair
Locations (2):
- United States (2):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Gorse GJ, McElrath MJ, Matthews TJ, Hsieh RH, Belshe RB, Corey L, Frey SE, Kennedy DJ, Walker MC, Eibl MM. Modulation of immunologic responses to HIV-1MN recombinant gp160 vaccine by dose and schedule of administration. National Institute of Allergy and Infectious Diseases AIDS Vaccine Evaluation Group. Vaccine. 1998 Mar;16(5):493-506. doi: 10.1016/s0264-410x(97)80003-5. PMID 9491504